CLINICAL TRIAL: NCT04849793
Title: The Effect of Acupressure on the Anxiety Level of Senior Nursing Students in the COVID-19 Pandemic
Brief Title: The Effect of Acupressure on the Anxiety Level
Acronym: Acupres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUniversity
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Anxiety
Keywords: Acupressure; Nursing students; Anxiety; COVID-19
MeSH Terms: conditions — Anxiety Disorders; COVID-19 | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm randomized controlled clinical trial
Who Masked: Participant
Masking Description: First of all, the names of all students will be listed alphabetically for the selection of 196 nursing students in the research population and 52 nursing students who will be the sample. Numbers between 1-196 will be written in front of each student in the ordered student list. 52 nursing students will be determined by randomization created in computer environment by an independent researcher who is not included in the study. A total of 52 students in the sample group determined by randomization will be separated according to the A and B groups created by the same statistician in computer environment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Before the intervention, the students will be asked to rub the area around the area to be pressed for 20-30 seconds with their palms. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in the area of warming, relaxing and preparatory will be reduced and the tissue will be relieved. After rubbing, each individual's pain threshold level will be taken as a basis in order not to cause tissue damage. The students will be asked to press the designated point manually with their thumb, index or middle finger for 5 seconds with a depth of 1-1.5 cm, rest for 2 seconds and continue the practice for 2 minutes. In the study group, an average of 13 minutes will be applied to HT7, LI4 and EX-HN3 points (five points in total) for two minutes each. The nursing students participating in the research will be given a total of 12 acupressure intervention remotely, three days a week, for four weeks, at least two hours after dinner and when they are calmest.
  Interventions: Other: Acupressure
- Control (No Intervention): No intervention will be made to the control group, only the data will be collected at the same time as the study group.

INTERVENTIONS:
Other: Acupressure — Before starting the application, the students will be asked to rub the area around the area to be pressed for 20-30 seconds with their palms. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in the area of warming, relaxing and preparatory will be reduced and the tissue will be relieved. . The students will be asked to press the designated point manually with their thumb, index or middle finger for 5 seconds with a depth of 1-1.5 cm, rest for 2 seconds and continue the practice for 2 minutes
  Other Names: Acupress
  Arms: Experimental

SUMMARY:
This randomized controlled study evaluates the effect of acupressure application on the anxiety level of senior nursing students.The hypothesis of this study is that acupressure reduces anxiety levels.

DETAILED DESCRIPTION:
Methods: In the study, 52 senior nursing students were randomly assigned to the study and control groups. The study group (n = 26) included Shen Men, the 7th acupuncture point (HT7) of the heart meridian located between the ulna and pisiform bones on the radial side of the flexor carpi ulnaris tendon, EX-HN3 (Yintang) located in the middle of the beginning of both eyebrows and the thumb and the LI4 points located in the space between the index finger (between the 1st and 2nd metacarpal bones of the hand, in the middle of the 2nd metacarpal bone on the radial side) will be applied for an average of 10 minutes. No intervention will be made to the control group (n = 26). In order to avoid ethical problems, both groups will be given an informative training on acupressure and anxiety content at the end of the study. The primary outcome of the study is the effect of acupressure on the state anxiety level of senior nursing students. The secondary outcome of the study is the effect of acupressure on trait anxiety level in senior nursing students. The results will be collected before the acupressure and in the 4th week of the last intervention.

ELIGIBILITY:
Inclusion Criteria:

The experimental group criteria to be included in the study;

* To voluntarily agree to participate in the study (those who signed the Informed Volunteer Form),
* Not having physical problems that would prevent acupressure application to HT7 (wrist), LI4 (the point where the thumb and index finger meet) and EX-HN3 (the middle point of the right and left eye level),
* Not having experience with acupressure,
* Not using drugs that affect anxiety level (antidepressants, analgesics, beta adrenoreceptor antagonists, dopamine agonists, etc.),
* Not using alcohol and drugs,
* Not having access to the devices required for internet and online education,
* Not being diagnosed with COVID-19 during the study,
* Not having any psychiatric diagnosis.,

The control group criteria to be included in the study;

* To voluntarily agree to participate in the study (those who signed the Informed Volunteer Form),
* Not having experience with acupressure,
* Not using drugs that affect anxiety level (antidepressants, analgesics, beta adrenoreceptor antagonists, dopamine agonists, etc.),
* Not having access to the devices required for internet and online education,
* Not using alcohol and drugs,
* Not being diagnosed with COVID-19 during the study,
* Not having any psychiatric diagnosis

Exclusion Criteria:

The experimental group criteria not to be included in the study;

* Not accepting voluntarily to participate in the study (those who did not sign the Informed Volunteer Form),
* Having a physical problem that prevents acupressure application to HT7 (wrist), LI4 (the point where the thumb and index finger meet) and EX-HN3 (the middle point of the right and left eye level),
* To have an acupressure experience,
* Using drugs that affect anxiety level (antidepressants, analgesics, beta adrenoreceptor antagonists, dopamine agonists, etc.),
* Having access to the devices required for internet and online education,
* Using alcohol and substance,
* Being diagnosed with COVID-19 during the study,
* Any psychiatric diagnosis

The control group criteria not to be included in the study;

* Not accepting voluntarily to participate in the study (those who did not sign the Informed Volunteer Form),
* To have an acupressure experience,
* Using drugs that affect anxiety level (antidepressants, analgesics, beta adrenoreceptor antagonists, dopamine agonists, etc.),
* Having access to the devices required for internet and online education,
* Using alcohol and substance,
* Being diagnosed with COVID-19 during the study,
* Having any psychiatric diagnosis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from before implementation and 4th week of practice
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also high

SECONDARY OUTCOMES:
Anxiety evaluated using the Trait Anxiety Scale | Change from before implementation and 4th week of practice
  In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher trait anxiety scores indicate that anxiety level is also high.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ALTUN UĞRAŞ, Doctorate, Study Director — gulaltun@mersin.edu.tr; Seher GÜRDİL YILMAZ, Doctorate, Principal Investigator — shrgrdl@hotmail.com; Ahmet KARAMAN, Doctorate, Principal Investigator — ahmet.karaman@mersin.edu.tr; Canan KANAT, MASTER, Principal Investigator — canankanat@mersin.edu.tr
Locations (1):
- Turkey, Mersin University,, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No